CLINICAL TRIAL: NCT04932525
Title: Gustave Roussy Cancer Profiling
Acronym: STING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A03547-32; 2020/3196 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2021-06-01; First posted 2021-06-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor, Unspecified, Adult
Keywords: immunological profiling; targetable oncogenic aberration
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: The proportion of patients presenting at least one genomic alteration will be estimated in the eligible NGS population and reported using frequency and proportion. The 95% two-sided confidence limits (95%CI) will be provided for the estimated proportion (binomial law). In addition, counts, proportions and 95%CI will be reported for each individual genomic alteration.
  Survival data will be analysed by standard time-to-event survival techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- solid tumor or hematological malignancy (Experimental)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Blood and tumor samples for Genetic Profiling research

SUMMARY:
The objective of STING study is to perform high throughput molecular analysis (next generation sequencing +/- immunological profiling) to estimate the proportion of patients with cancer presenting at least one targetable genomic alteration.

DETAILED DESCRIPTION:
STING is a biology driven, multicenter study designed to identify actionable molecular alterations in cancer patients and to explore mechanisms of sensitivity and resistance to anti-cancer treatment

* In this trial, high throughput analysis will be carried out using next generation sequencing, and immunological profiling
* Patients included in the STING study and for whom a targetable genomic alteration had been identified might be subsequently included in a clinical trial running at Gustave Roussy or another participating center.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histology: solid malignant tumor or hematological malignancy.
3. Patient with a social security in compliance with the French law relating to biomedical research (Article L.1121-11 of French Public Health Code)
4. Voluntary signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

1. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in a clinical trial or which would jeopardize compliance with the protocol
2. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
3. Pregnant or breast-feeding women
4. Minors (Age < 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2033-05-10 (Estimated); Study Completion 2033-05-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients presenting at least one targetable genomic alteration | 2 months after the last enrollment
  Number of patients presenting at least one targetable genomic alteration
Proportion of patients presenting at least one targetable genomic alteration | 2 months after the last enrollment
  Proportion of patients presenting at least one targetable genomic alteration

SECONDARY OUTCOMES:
Rate of molecular profiling information including utilization of information for standard regimens or clinical trials of molecularly targeted therapies | 2 months after the last enrollment
  For a patient with molecular results available utilization of molecular profiling information is defined as Inclusion in a clinical trial assessing a drug matched to the molecular alteration And/or Treatment with an approved drug matched with the molecular alteration
Objective response rate | 24 months post treatment after the last enrollment
Progression-free survival | 24 months post treatment after the last enrollment
Overall survival | 24 months post treatment after the last enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, MD PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (4):
- France (4):
  - Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne
  - Hôpital Marie-Lannelongue, Le Plessis-Robinson
  - Hôpital Saint-Joseph, Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Derived] Rodriguez J, Baldini C, Bayle A, Pages A, Danlos FX, Vasseur D, Rouleau E, Lacroix L, Alonso de Castro B, Goldschmidt V, Seknazi L, Hollebecque A, Michot JM, Champiat S, Marabelle A, Ouali K, Marzac C, Ponce S, Micol JB, Chaput N, Massard C, Italiano A. Impact of Clonal Hematopoiesis-Associated Mutations in Phase I Patients Treated for Solid Tumors: An Analysis of the STING Trial. JCO Precis Oncol. 2024 May;8:e2300631. doi: 10.1200/PO.23.00631. PMID 38815178
- [Derived] Helal C, Pobel C, Bayle A, Vasseur D, Nicotra C, Blanc-Durand F, Naoun N, Bernard-Tessier A, Patrikidou A, Colomba E, Flippot R, Fuerea A, Auger N, Ngo Camus M, Besse B, Lacroix L, Rouleau E, Ponce S, Italiano A, Loriot Y. Clinical utility of plasma ctDNA sequencing in metastatic urothelial cancer. Eur J Cancer. 2023 Dec;195:113368. doi: 10.1016/j.ejca.2023.113368. Epub 2023 Oct 6. PMID 37897866
- [Derived] Aldea M, Tagliamento M, Bayle A, Vasseur D, Verge V, Marinello A, Danlos FX, Blanc-Durand F, Bernard E, Cerbone L, Mosele MF, Renneville A, Hadoux J, Loriot Y, Sakkal M, Vozy A, Sarkozy C, Smolenschi C, Nicotra C, Martin-Romano P, Boccon-Gibod C, Habza W, Lazarovici J, Ponce S, Hollebecque A, Marzac C, Lacroix L, Barlesi F, Andre F, Besse B, Rouleau E, Italiano A, Micol JB. Liquid Biopsies for Circulating Tumor DNA Detection May Reveal Occult Hematologic Malignancies in Patients With Solid Tumors. JCO Precis Oncol. 2023 Mar;7:e2200583. doi: 10.1200/PO.22.00583. PMID 36862966